CLINICAL TRIAL: NCT02021994
Title: BPM Cuff： 15-24cm, 20-34cm, 30-44cm, 40-48cm, 22-42cm
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 9
Record Dates: First submitted 2013-09-10; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Blood Pressure

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Arm Automatic Electronic BPM
- mercury sphygmomanometer

SUMMARY:
The purpose of this study is to verify the accuracy of the 5 blood pressure cuffs, with blood pressure monitor device.

The cuff range is as follows:

15cm-24cm, 20cm-34cm, 30cm-44cm, 40cm-48cm, and 22cm-42cm

ELIGIBILITY:
Inclusion Criteria:

1. Normal adult or adults with Hypertension

   Exclusion Criteria:

   ⎯1) people with serious arrhythmia
2. Patients with Takayasu arteritis
3. people wit adverse vascular peripheral circulation
4. people with upper limbs vein thrombosis
5. people who is weak

Ages: 20 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: resident of a community
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
All the test results of the electronic blood pressure monitor with 5 cuffs is within the accuracy creteria, with the mercury sphygmomanometer as control | 1 day